CLINICAL TRIAL: NCT05967442
Title: A Randomized, Placebo-Controlled, Double-Blind Study of the Effects of Magnesium Compared to Conventional Therapy on Acute Migraine
Brief Title: Magnesium Versus Prochlorperazine Versus Metoclopramide for Migraines
Acronym: MAGraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AHC-7192-D5000322
Record Dates: First submitted 2020-01-09; First posted 2023-08-01 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Migraine; Headache
Keywords: magnesium; migraine; headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Magnesium Sulfate; Metoclopramide; Prochlorperazine; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Magnesium (Experimental): Magnesium Sulfate 2gm in 50ml D5W over 20 minutes
  Interventions: Drug: Magnesium Sulfate
- Metoclopramide (Active Comparator): Metoclopramide 10mg in 50ml D5W over 20 minutes
  Interventions: Drug: Metoclopramide 10mg
- Prochlorperazine (Active Comparator): Prochlorperazine in 50ml D5W over 20 minutes
  Interventions: Drug: Prochlorperazine (Compazine) Injection

INTERVENTIONS:
Drug: Magnesium Sulfate — Magnesium Sulfate 2gm in 50ml D5W over 20 minutes
  Arms: Magnesium
Drug: Metoclopramide 10mg — Metoclopramide 10mg in 50ml D5W over 20 minutes
  Arms: Metoclopramide
Drug: Prochlorperazine (Compazine) Injection — Prochlorperazine 10mg in 50ml D5W over 20 minutes
  Arms: Prochlorperazine

SUMMARY:
This investigation describes a proposed clinical trial that will evaluate the relative efficacy of intravenous magnesium sulfate for the treatment of migraine compared to intravenous metoclopramide (Reglan) and intravenous prochlorperazine (Compazine) in the treatment of acute headache and migraine in adult patients. The ultimate objective will be clinical application of these drugs in the emergency department for the treatment of acute headache and migraine.

The two phenothiazines (metoclopramide and prochlorperazine) have been routinely utilized in the treatment of acute headache and migraine in the emergency department setting. Per the 2017 American Headache Society guidelines, both intravenous metoclopramide and intravenous procholorperazine are recommended as "clinicians should offer" agents with level B evidence. Of note, there are no agents with level A evidence purported by this guideline for acute management of migraine. The same guideline offers "no recommendation can be made regarding the role of intravenous magnesium for adults who present to the ED with acute migraine. However intravenous magnesium may be of benefit to patients who present with migraine with aura." Multiple trials have evaluated intravenous magnesium's safety and efficacy in the management of acute migraine. These have demonstrated the tolerability of intravenous magnesium on a with breadth of patients. Most commonly the primary adverse event was flushing which self-resolved. No cases of hypotension were reported.

None of these study agents have been withdrawn from the market.

DETAILED DESCRIPTION:
Migraine or severe headache affected one-fifth of women and one-tenth of men in 2015 and is one of the leading causes of disability in the world. Over one million visits to emergency departments (ED) in the US are due to migraines. Migraine, previously believed to be a vascular disorder, is caused by inflammation due to vasodilation in the meninges secondary to the release of vasoactive neuropeptides by stimulation of the trigeminal nerve. This inflammation can result in symptoms such as headache, nausea, vomiting, dizziness, photophobia and phonophobia.

Despite migraine being a common disorder, there has yet to be a cure. Several classes of medications have been studied for the treatment of migraine. Recently, conventional therapy has shifted to the use of antidopaminergics including prochlorperazine, metoclopramide and haloperidol, nonsteroidal anti-inflammatory drugs (NSAIDs) such as ibuprofen and naproxen, and triptans, sumatriptan being the most commonly utilized. 5Although intravenous opioids have historically been the most common treatment for migraines, their use has fallen out of favor due to their association with increased recurrence of headaches and ED visits, abuse potential, and most recently severe intravenous opiate shortage. Alternative treatments include ketamine, propofol, dihydroergotamine and magnesium.

Magnesium is an intracellular cation that has been associated with both the function of serotonin and regulation of vascular tone, which are both mechanisms that implicate its role in the treatment of migraine. Intravenous magnesium sulfate has been studied as a treatment for migraine compared to placebo, metoclopramide and prochlorperazine. These studies have shown that magnesium is well-tolerated with a good safety profile and may be efficacious in the treatment of migraine. Metoclopramide, prochlorperazine and magnesium have been recommended in clinical practice guidelines and have become routine standard of care for treatment of migraine in this emergency department. However, no trial has evaluated these modalities simultaneously in the same population. The purpose of our study is to compare the relative efficacy for magnesium, metoclopramide, and prochlorperazine in the treatment of headache and migraine.

Via monthly block randomization, patients will be given one of three guideline recommended study drugs. Allocation will be concealed by a pharmacist (not participating in the rest of the study) solely designated to choose which drug will be the assigned study drug for each month. The pharmacists, physicians, and nurses participating in administration of the medications will be blinded to which drug is being administered during each month. Metoclopramide, prochlorperazine and magnesium have been recommended in clinical practice guidelines and have become routine standard of care for treatment of migraine in this emergency department. All three study drugs will be stored in the investigational medication refrigerator located in the main pharmacy. A pharmacist on duty in the emergency department will obtain the medication from the refrigerator and deliver it to the bedside nurse who is actively caring for the patient after an order from the physician.

The primary outcome of this study will be mean change in pain from baseline to 30 minutes after initiation of infusion (as defined on a 11-point Numeric Rating Scale. Secondary endpoints include mean change in pain from baseline to 60 minutes and 120 minutes after initiation of infusion (as defined on a 11-point Numeric Rating Scale), time to emergency department discharge, and adverse effects due to administration of study drug (hypotension, flushing, akathisia, dystonia, nausea, vomiting, dizziness, drowsiness, other self-reported adverse effects).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years or older
* Able to provide informed consent
* Primary diagnosis of headache or migraine
* Between October 1, 2018 to April 1, 2020
* Presenting to Advocate Christ Medical Center emergency department and meet clinical assessment per physician

Exclusion Criteria:

* Pregnancy defined as a positive urine HCG
* Stated history of renal impairment
* Allergy or sensitivity to any study drugs
* Concomitant treatment at the time of study drug administered in the emergency department
* Patients with a history of this study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2023-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Cirone, MD, Principal Investigator — advocate christ medical center
Locations (1):
- Advocate Christ Medical Center, Oak Lawn, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Magnesium | Metoclopramide | Prochlorperazine
Started | 61 | 44 | 52
Completed | 61 | 44 | 52
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Magnesium | Metoclopramide | Prochlorperazine | Total
Number analyzed (Participants) | 61 | 44 | 52 | 157
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34 [27 to 48] | 37.5 [29.5 to 48] | 37.5 [27 to 47.5] | 36 [27 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 33 | 46 | 123
  Male | 17 | 11 | 6 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 9 | 20
  Not Hispanic or Latino | 55 | 39 | 42 | 136
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: 30 Minute Pain Score
Description: Scores range from 0-10. A higher score, denotes more pain
Time Frame: 30 minutes after initiation
Population: Full cohort
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Magnesium | Metoclopramide | Prochlorperazine
Number analyzed (Participants) | 61 | 44 | 52
score on a scale | 3 [1 to 4] | 3 [1 to 4] | 3 [1 to 5]

2. Secondary Outcome: Length of Stay
Description: Emergency Department Length of stay. Measured from time of arrival to time of discharged documented in the electronic medical record.
Time Frame: From time of arrival to time of discharge.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Magnesium | Metoclopramide | Prochlorperazine
Number analyzed (Participants) | 61 | 44 | 52
minutes | 325 [274 to 410] | 308 [263.5 to 403] | 332 [268.5 to 391]

3. Secondary Outcome: Need for Rescue Analgesia
Description: Percentage of participants who had necessity for rescue analgesics after study drug administration
Time Frame: From time of arrival to time of discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Magnesium | Metoclopramide | Prochlorperazine
Number analyzed (Participants) | 61 | 44 | 52
Participants | 26 | 15 | 17

ADVERSE EVENTS:
Time Frame: Adverse effects were investigated at every VAS evaluation time time point, 30 minutes, 60 minutes, and 120 minutes.
Description: Due to the isolated time frame of observation and the established safety profile of these medications, no patients were at risk for all-cause mortality.
Arm/Group | Magnesium | Metoclopramide | Prochlorperazine
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/44 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/44 | 0/52
Other Adverse Events (participants affected / at risk) | 0/61 | 0/44 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT05967442/Prot_SAP_002.pdf